CLINICAL TRIAL: NCT01557231
Title: Epidemiology of OA Pain
Brief Title: Epidemiology of Osteoarthritis (OA) Pain
Status: Completed | Type: Observational
Sponsor: Northwestern University (Other)
Collaborators: ZARS Pharma Inc. (Industry)
Responsible Party: Principal Investigator, Thomas J. Schnitzer, Professor, Northwestern University
Other Study IDs: STU00059872
Record Dates: First submitted 2012-03-14; First posted 2012-03-19 (Estimated); Last update posted 2018-03-29 (Actual); Status verified 2018-03

CONDITIONS: Osteoarthritis
Keywords: OA; osteoarthritis; pain; variability; activity; treatment
MeSH Terms: conditions — Osteoarthritis; Pain; Motor Activity

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- No treatment: OA

SUMMARY:
Chronic pain, by definition, persists over long periods of time, but both sufferers of pain and their caregivers are aware that pain levels can fluctuate greatly over time. Being able to define pain variability and its underlying causes would be an important advance in our understanding of chronic pain, and would in turn lead to better approaches to the treatment of chronic pain. In this study, the investigators propose to evaluate in 60 people with chronic pain of the knee due to osteoarthritis over 3 months, collecting data regarding magnitude of pain, physical activity level, and medication status twice daily during this period of time. The investigators then will assess the variability in pain levels over time, the frequency of "flares" of osteoarthritis (OA) pain and their relationship to physical activity, medications, and clinical descriptors of the population, e.g., age, gender, body mass index (BMI). Additionally, evaluations will be made regarding temporal patterns of OA knee pain as well as assessment of subgroups of patients with the overall group being studied.

ELIGIBILITY:
Inclusion Criteria:

1. Men and women, age 40 years and above
2. Knee pain most days of the week for the past month
3. Diagnosis of knee OA
4. Meet ACR criteria for knee OA
5. No significant limitations in physical activity
6. Own and able to use a cellular phone capable of text messaging
7. Able to return for all clinic visits
8. Able to read and understand the informed consent document

Exclusion Criteria:

1. Use of a walker to ambulate or inability to ambulate (use of cane is allowed)
2. Other forms of arthritis
3. Other major causes of pain that could be expected to interfere with assessment of pain during this trial, e.g., recurrent migraine, back pain, fibromyalgia
4. Scheduled for and likely to need joint replacement surgery in the next 3 months
5. Any medical condition that in the judgment of the investigator would make the participant not suitable for the study
6. Living in a long-term care facility

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Individuals with OA
Sampling Method: Non-Probability Sample
Enrollment: 86 (Actual)
Dates: Start 2012-03; Primary Completion 2015-09 (Actual); Study Completion 2015-09 (Actual)

PRIMARY OUTCOMES:
pain magnitude | 6 months
  magnitude of pain will be evaluated 3x/day

SECONDARY OUTCOMES:
self-reported activity level | 6 months
  data will be collected 3x/day; Likert 1-5 scale

CONTACTS AND LOCATIONS:
Locations (1):
- Northwestern University Feinberg School of Medicine, Chicago, Illinois, United States